CLINICAL TRIAL: NCT05603065
Title: A Randomized, Open-label, Uncontrolled Study of Tislelizumab in Combination With Chemotherapy or Radiation Therapy for Neoadjuvant Therapy for Resectable Thoracic Esophageal Squamous Cell Carcinoma (TINES)
Brief Title: Tislelizumab With Chemotherapy or Radiation for Neoadjuvant Therapy of Esophageal Squamous Cell Carcinoma (TINES)
Acronym: TINES
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No. XJTU1AF2022LSK-374
Record Dates: First submitted 2022-10-20; First posted 2022-11-02 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2022-10

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Tislelizumab; Neoadjuvant therapy; Immunotherapy; Esophageal squamous cell carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — tislelizumab; Cisplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Cohort study
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy (Active Comparator)
  Interventions: Drug: Tislelizumab + cisplatin + paclitaxel
- Radiotherapy (Active Comparator)
  Interventions: Drug: Tislelizumab + radiotherapy

INTERVENTIONS:
Drug: Tislelizumab + cisplatin + paclitaxel — Tislelizumab 200mgD1 + cisplatin 75mg/m^2D1 + paclitaxel 150mg/m^2D1 Q3W 3 cycles
  Arms: Chemotherapy
Drug: Tislelizumab + radiotherapy — Tislelizumab 200mgQ3W 3 cycles + radiotherapy (23 times in total, 1.8 Gy per dose, 5 times a week)
  Arms: Radiotherapy

SUMMARY:
Esophageal squamous cell carcinoma (ESCC), one of the most common subtypes of esophageal cancer, has a poor prognosis and low 5-year overall survival. At present, the treatment of ESCC includes chemotherapy, immunity, radiotherapy, surgery and other methods, and in recent years, the treatment regimen of immune combined chemotherapy has begun to show results in the treatment of esophageal cancer. Tislelizumab has demonstrated good efficacy in advanced esophageal cancer and in the second- and third-line treatment. At present, neoadjuvant immunization is carried out less, and neoadjuvant immunization plus chemoradiotherapy has been achieved With a pCR rate of 55.6 and AEs of grade III and above 65%, and studies have shown that radiotherapy has immunosensitizing and coordinating effects, whether immunotherapy combined with radiotherapy has a better efficacy is worth further investigation. This review intends to conduct a randomized, open-label, uncontrolled study of tislelizumab in combination with chemotherapy or radiation therapy for neoadjuvant therapy for resectable locally advanced thoracic esophageal squamous cell carcinoma with a view to providing a new option for resectable locally advanced ESCC.

ELIGIBILITY:
Inclusion Criteria:

* (1) The subjects voluntarily joined the study and signed the informed consent form, with good compliance and follow-up;
* (2) 18 years old≤ age≤ 79 years old, male or female;
* (3) ECOG score 0~1 points;
* (4) Patients with pathological (histological or cytology) confirmed esophageal squaf cell carcinoma; According to the eighth edition of the clinical tumor TNM stage, subjects were resectable cT2-4aNanyM0;
* (5) Have measurable lesions (according to RECIST 1.1 criteria, tumor lesion CT scan length diameter≥ 10mm lymph node lesion CT scan short diameter ≥15mm);
* (6) Those who were first diagnosed with esophageal squamous cell carcinoma before enrollment and did not undergo radiotherapy, chemotherapy, immunity, surgery and targeted therapy;
* (7) Able to eat a liquid diet or above, no signs before esophageal perforation or esophageal ulcers, and able to tolerate surgery;
* (8) The main organs function normally, that is, meet the following standards:

  1. Routine blood examination must be consistent (no blood transfusion, no hematopoietic factor and no correction with drugs within 14 days): ANC≥1.5×109/L; PLT≥100×109；HB≥90g/L；
  2. Biochemical tests must meet the following standards: TBIL≤1.5×ULN; ALT、AST≤2.5×ULN； serum creatinine sCr≤1.5×ULN, endogenous creatinine clearance≥50mL/min (Cockcroft-Gault formula); ALB≥30g/L；
  3. The coagulation function must meet: INR≤1.5×ULN and APTT≤1.5×ULN;
  4. Normal or mild to moderate lung function and can tolerate esophageal cancer surgery. Preoperative lung function examination should meet: VC% > 60%; FEV1 > 1.2 L，FEV1% > 40%； DLco>40%。

Exclusion Criteria:

* (1) Have any active autoimmune disease or history of autoimmune disease (as follows, but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (may be included after hormone replacement therapy)); Patients with vitiligo or childhood asthma that have been in complete remission and do not require any intervention in adulthood are excluded, but patients requiring medical intervention with bronchodilators are not included;
* (2) Patients with congenital or acquired immunodeficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B, hepatitis C or co-infection with hepatitis B and C;
* (3) immunosuppressive drugs have been used within 14 days prior to first use of study drug, excluding nasal and inhaled corticosteroids or physiologic doses of systemic steroids (i.e., not more than 10mg/day prednisone or its equivalent);
* (4) The patient lost ≥ 10% body weight within 6 months before enrollment, or the BMI < 18.5kg/m2, or PG-SGA reached grade C;
* (5) Live attenuated vaccine within 4 weeks prior to the first dose or planned for the duration of the study;
* (6) other malignant tumors in the past 3 years;
* (7) uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg, despite optimal medical therapy); Patients with a new diagnosis of angina within 3 months prior to screening or myocardial infarction events within 6 months prior to screening; Arrhythmias (including QTcF: ≥450ms for men and 470ms ≥ women) require long-term use of antiarrhythmic drugs and grade II cardiac insufficiency ≥ New York Heart Association;
* (8) Those with a history of severe lung or heart disease;
* (9) Complicated by severe infection (eg, requiring intravenous antibiotics, antifungal or antiviral drugs) within 4 weeks before the first dose, or unexplained fever >38.5°C during screening/before the first dose;
* (10) Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* (11) Pregnant or lactating women; Patients of childbearing potential who are unwilling or unable to use effective contraception;
* (12) Known allergic reactions, hypersensitivity reactions or intolerances to investigational drugs and their excipients;
* (13) Subjects who are participating in other clinical studies or whose first dose is less than 4 weeks from the end of the previous clinical study (last dose), or who have 5 half-lives of the study drug;
* (14) Subject has a known history of psychotropic substance abuse, alcohol or drug abuse;
* (15) Any condition that the investigator believes is likely to harm the subject or cause the subject to be unable to meet or perform the study requirements;
* (16) After neoadjuvant therapy, the patient cannot tolerate surgery or is not suitable for surgery due to the progression of the disease.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | From date of randomization until the date of first documented progression or date of death from any cause whichever came first, up to 100 weeks
  postoperative pathological examination shows no carcinological tissue residue

SECONDARY OUTCOMES:
Primary pathologic response rate (MPR) | From date of randomization until the date of first documented progression or date of death from any cause whichever came first, up to 100 weeks
  postoperative pathological examination shows a residual < of 10% of cancerous tissue
Objective response rate (ORR) of primary lesions (RECIST v1.1) | From date of randomization until the date of first documented progression or date of death from any cause whichever came first, up to 100 weeks
  the proportion of patients whose tumors shrink to a certain amount and remain for a certain period of time under imaging measurements, including complete response (CR, Complete Response) and partial response (PR, partial response) cases CR is defined as the complete disappearance of all target lesions except nodular disease. All target nodules must be reduced to normal size (minor axis< 10 mm). All target lesions must be evaluated.
  PR is defined as the sum of the diameters of all measurable target lesions less than 30% ≥ baseline. The target nodule is summed and the short diameter is used, while all other target lesions are combined and the longest diameter is used. All target lesions must be evaluated.
Disease-free survival (DFS) | From date of randomization until the date of first documented progression or date of death from any cause whichever came first, up to 100 weeks
  the time between postoperative surgery and recurrence of disease or death (for any cause)
Over all survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause whichever came first, up to 100 weeks
  the time from postoperative surgery to death (for any reason)
Safety in the neoadjuvant phase and postoperative phase | From date of randomization until the date of first documented progression or date of death from any cause whichever came first, up to 100 weeks
  according to the Common Acute and Subacute Toxicity Grading Standard (CTCAE 5.0), the adverse reactions after each immune combined radiotherapy or immune combined chemotherapy in the neoadjuvant therapy stage and the postoperative adverse reactions were evaluated
Quality of life measurement and evaluation 1 | From date of randomization until the date of first documented progression or date of death from any cause whichever came first, up to 100 weeks
  according to the QLQ-C30 scale of the Quality of Life Survey, the quality of life after neoadjuvant therapy was assessed
Quality of life measurement and evaluation 2 | From date of randomization until the date of first documented progression or date of death from any cause whichever came first, up to 100 weeks
  according to the QLQ-OES18 special scale for esophageal cancer, the quality of life after neoadjuvant therapy was assessed

CONTACTS AND LOCATIONS:
Overall Officials: Junke Fu, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No